CLINICAL TRIAL: NCT03888599
Title: Knowledge and Attitudes Towards Human Papillomavirus Infections and HPV Vaccination Among Undergraduate Health Students From Switzerland
Brief Title: Knowledge and Attitudes Towards Human Papillomavirus Infections and HPV Vaccination
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jeannot Emilien, Principal Investigator, University Hospital, Geneva
Other Study IDs: Req-2019-00118
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: HPV-Related Cervical Carcinoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: knowledge questioannaire — , all enrolled undergraduate student received directly on your email the online questionnaire based on the "Fluid Survey tool", which was an on line survey tool (https://fluidsurveys.com/)

SUMMARY:
A better understanding of the target audiences about HPV infection and HPV vaccination would surely allow for a better spread of this vaccination in Switzerland. In order to know if the target audiences are properly informed, we have decided to carry out a study evaluating their level of knowledge on a particular audience that are the men and women undergraduate nurse.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women and men aged between 18-36 years
* Understands study procedures and accepts voluntarily to participle of the study

Exclusion Criteria:

.Don't understand french language

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women above the age of 18 years, currently attending the School of Health Sciences of three selected Swiss towns to obtain a nurse or midwife degree
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire about basic knowledge HPV infection | 3 months
  Percentage of right answer of the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Jeannot, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided